CLINICAL TRIAL: NCT00853021
Title: Phase II Open Label Trial of rIL-2 and Bevacizumab Combination in Patients With Metastatic Clear Cell Renal Carcinoma
Brief Title: Bevacizumab and Aldesleukin in Treating Patients With Metastatic Clear Cell Carcinoma of the Kidney
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jorge A. Garcia, MD (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Jorge A. Garcia, MD, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE8804; P30CA043703 (NIH); CASE8804 (Other: Case Comprehensive Cancer Center); 7493 (Other: Cleveland Clinic IRB)
Record Dates: First submitted 2009-02-26; First posted 2009-02-27 (Estimated); Results first posted 2015-08-24 (Estimated); Last update posted 2019-06-05 (Actual); Status verified 2019-05

CONDITIONS: Kidney Cancer
Keywords: clear cell renal cell carcinoma; recurrent renal cell cancer; stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — aldesleukin; chiron; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab and Aldesleukin (Experimental)
  Interventions: Biological: aldesleukin; Biological: bevacizumab

INTERVENTIONS:
Biological: aldesleukin — SQ Aldesleukin (Days 1-5) Monday through Friday for six weeks followed by a two-week break.
  Other Names: rIL-2 (NSC3773364); Proleukin®; Chiron
Biological: bevacizumab — Bevacizumab will be administered on day -14, then on day 1 and every 2 weeks thereafter (days 1, 15, 29, and 42) in a continuous manner.

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Biological therapies, such as aldesleukin, may stimulate the immune system in different ways and stop tumor cells from growing. Giving bevacizumab together with aldesleukin may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving bevacizumab together with aldesleukin works in treating patients with metastatic clear cell carcinoma of the kidney.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the effect of the combination of bevacizumab and aldesleukin on progression-free survival of patients with good- or intermediate-risk metastatic clear cell renal cell carcinoma.

Secondary

* To determine the objective response rate in patients receiving this regimen.
* To determine the time to progression in patients receiving this regimen.
* To evaluate immunomodulatory effects of this regimen in patients
* To evaluate the toxicity of this regimen in these patients.

OUTLINE: Patients receive bevacizumab IV over 30-90 minutes on days -14, 1, 15, 29, and 42 and aldesleukin subcutaneously on days 1-5, 8-12, 15-19, 22-26, 29-33, and 36-40. Courses repeat every 8 weeks for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients achieving complete response after completion of study therapy may receive 1 additional course of therapy.

After completion of study therapy, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed renal cell carcinoma (RCC) of clear cell histology with or without sarcomatoid features

  * Metastatic disease
  * No non-clear cell RCC (i.e., papillary, collecting-duct, or chromophobe)
* Good- or intermediate-risk category as defined by having ≤ 2 of the following factors:

  * No prior nephrectomy
  * Karnofsky performance status < 80%
  * Hemoglobin < 12 g/dL
  * Corrected calcium > 10.0 mg/dL
  * LDH > 1.5 times upper limit of normal (ULN)
* Must have undergone a nephrectomy at least 28 days ago
* Measurable or evaluable disease by RECIST
* No significant effusions and/or ascites
* No prior or concurrent brain or CNS metastasis

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy of ≥ 3 months
* WBC ≥ 3,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9.5 g/dL
* Creatinine ≤ 2.0 mg/dL
* Total bilirubin ≤ 1.5 mg/dL
* AST ≤ 5.0 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN (≤ 10 times ULN with bone metastasis)
* Calcium ≤ 12 mg/dL
* Urine protein:creatinine ratio ≤ 1.0
* INR ≤ 1.5 (unless receiving warfarin therapy)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No uncontrolled seizure disorder
* No known HIV positivity
* No local or systemic infections requiring IV antibiotics within the past 28 days
* No significant traumatic injury in the past 28 days
* No serious non-healing wound, ulcer, or acute bone fracture
* No evidence of bleeding diathesis or coagulopathy
* No other malignancy except basal cell or squamous cell carcinoma of the skin, carcinoma in-situ of the uterine cervix, or any malignancy treated with curative intent and in complete remission for > 3 years
* No history of serious systemic or severe cardiovascular disease, including any of the following:

  * Arterial thromboembolic event (including transient ischemic attack)
  * Cerebrovascular accident
  * Unstable angina
  * Myocardial infarction within the past 6 months
  * Uncontrolled hypertension (BP > 160/110 mm Hg on medication)
  * Uncontrolled cardiac arrhythmia
  * Congestive heart failure
  * Angina pectoris
  * NYHA class III-IV cardiovascular disease
  * Peripheral vascular disease ≥ grade II
* No history of abdominal fistula and/or bowel or gastric perforation within the past 6 months
* No history of other diseases, metabolic dysfunction, or physical or laboratory examination findings giving reasonable suspicion of a disease or condition that contraindicate the use of investigational drugs, or that might affect the interpretation of study results, or that render patient at high-risk for treatment complications

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior organ allografts
* No prior systemic therapy for metastatic clear cell renal cell carcinoma
* At least 4 weeks since prior radiotherapy and recovered

  * Radiotherapy for control of pain from skeletal lesions allowed within the past 28 days
* More than 12 months since prior adjuvant therapy
* More than 7 days since prior fine-needle aspirations or core biopsies
* More than 28 days since prior and no concurrent major surgery requiring general anesthesia or open biopsy
* No concurrent aspirin, corticosteroids (except at replacement doses), barbiturates, or other investigational agents

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2005-12; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge A. Garcia, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bevacizumab and Aldesleukin
Started | 26
Completed | 21
Not Completed | 5
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 2
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab and Aldesleukin
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 25
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression free survival is defined as the time between registration and progression of disease as defined by the RECIST criteria where there is a 20% increase in the diameter of the tumor and at least a 5mm absolute increase in diameter.
Time Frame: From baseline (day -14) to disease progression (reported at 2 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab and Aldesleukin
Number analyzed (Participants) | 26
months | 9.6 [4.1 to 16.9]

2. Secondary Outcome: Objective Response Rate (Complete and Partial Response)
Description: Objective response rate to be assigned a status of PR or CR per RECIST criteria, with Complete Response (CR) referring to the disappearance of all target lesions, Partial Response (PR) referring to at least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD.
  Changes in tumor measurements must be confirmed by repeat assessments that should be performed no less than 4 weeks after the criteria for response are first met.
Time Frame: 4 weeks after end of treatment
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab and Aldesleukin
Number analyzed (Participants) | 26
percentage of participants | 15

3. Secondary Outcome: Percentage of Patients With Constitutional Adverse Events
Description: Toxicity Criteria: The NCI graded common clinical toxicity scale (NCI Version 2.0) will be employed to grade observed toxicity of fatigue and fever/chills
Time Frame: From start of treatment to 30 days after treatment
Measure: Number; unit: percentage of patients
Arm/Group | Bevacizumab and Aldesleukin
Number analyzed (Participants) | 26
percentage of patients | 42

4. Secondary Outcome: Percentage of Patients With Neutropenia
Description: Toxicity Criteria: The NCI graded common clinical toxicity scale (NCI Version 2.0) will be employed to grade observed toxicity of neutropenia
Time Frame: From start of treatment to 30 days after treatment
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab and Aldesleukin
Number analyzed (Participants) | 26
percentage of participants | 12

5. Other Pre Specified Outcome: Peripheral Blood CD1c+ Myeloid Dendritic Cells
Description: Peripheral blood mononuclear cells (PBMC) and plasma were separated by centrifugation. Targeted cells were isolated by a magnetic labeling system. Total RNA was isolated and then amplified by (Polymerase Chain Reactions) PCR to measure levels of the immune parameter.
Time Frame: Baseline (day -14), Beginning and end of cycle 1 (day 1, 57)
Reporting Status: Not Posted

6. Other Pre Specified Outcome: CD303+ Plasmacytoid Dendritic Cells
Description: as for outcome 5
Time Frame: Baseline (day -14), beginning and end of cycle 1 (day 1, 57)
Reporting Status: Not Posted

7. Other Pre Specified Outcome: IL-8 Levels
Description: as for outcome 5
Time Frame: Baseline (day -14), beginning and end of cycle 1 (day 1, 57)
Reporting Status: Not Posted

8. Other Pre Specified Outcome: CD4+ Treg Cells
Description: as for outcome 5
Time Frame: Baseline (day -14), beginning and end of cycle 1 (day 1, 57)
Reporting Status: Not Posted

9. Other Pre Specified Outcome: CD25+ Treg Cells
Description: as for outcome 5
Time Frame: Baseline (day -14), beginning and end of cycle 1 (day 1, 57)
Reporting Status: Not Posted

10. Other Pre Specified Outcome: T-helper Cells (Type 1,2)
Description: as for outcome 5
Time Frame: Baseline (day -14), beginning and end of cycle 1 (day 1, 57)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 18 Months
Description: From beginning of treatment to 30 days after treatment. The maximum time was 18 months
Arm/Group | Bevacizumab and Aldesleukin
Serious Adverse Events (participants affected / at risk) | 9/26
Other Adverse Events (participants affected / at risk) | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab and Aldesleukin (N=26)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Abdominal pain or cramping (Gastrointestinal disorders) | 1 (2)
Ascites (Gastrointestinal disorders) | 1 (1)
Heart failure (Cardiac disorders) | 2 (2)
Confusion (Psychiatric disorders) | 1 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Infection without neutropenia (Infections and infestations) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab and Aldesleukin (N=26)
Abdominal pain or cramping (Gastrointestinal disorders) | 6 (11)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Respiratory, thoracic and mediastinal disorders) | 13 (27)
Anorexia (Gastrointestinal disorders) | 21 (49)
Arthralgia (joint pain) (Musculoskeletal and connective tissue disorders) | 7 (15)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (4)
Constipation (Gastrointestinal disorders) | 8 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (14)
Creatinine Increased (Investigations) | 2 (2)
Dehydration (Gastrointestinal disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 18 (32)
Dizziness/lightheadedness (Nervous system disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 8 (9)
Dyspepsia (Gastrointestinal disorders) | 4 (6)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 11 (19)
Edema (General disorders) | 2 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Fatigue (lethargy, malaise, asthenia) (General disorders) | 26 (108)
Fever (in the absence of neutropenia, where neutropenia is defined as AGC<1.0 x 10e9/L) (General disorders) | 18 (44)
abdominal bloating (Gastrointestinal disorders) | 3 (5)
acid reflux (Gastrointestinal disorders) | 4 (4)
vomiting (Gastrointestinal disorders) | 12 (25)
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 2 (3)
Headache (Nervous system disorders) | 8 (11)
Hematuria (in the absence of vaginal bleeding) (Renal and urinary disorders) | 2 (6)
anemia (Blood and lymphatic system disorders) | 4 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (5)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (5)
Hypertension (Vascular disorders) | 6 (13)
Hypotension (Vascular disorders) | 3 (3)
Injection site reaction (General disorders) | 20 (53)
Insomnia (Psychiatric disorders) | 9 (11)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2)
Lymphopenia (Investigations) | 2 (2)
Mood alteration-anxiety, agitation (Psychiatric disorders) | 4 (8)
Mood alteration-depression (Psychiatric disorders) | 4 (4)
Mouth dryness (Gastrointestinal disorders) | 2 (5)
Muscle weakness (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 2 (3)
Myalgia (muscle pain) (Musculoskeletal and connective tissue disorders) | 12 (14)
Nausea (Gastrointestinal disorders) | 22 (70)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 3 (4)
Pain (General disorders) | 10 (19)
Proteinuria (Renal and urinary disorders) | 3 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 5 (8)
Rigors, chills (General disorders) | 26 (71)
Stomatitis/pharyngitis (oral/pharyngeal mucositis) (Infections and infestations) | 12 (24)
Sweating (diaphoresis) (General disorders) | 3 (6)
Syncope (fainting) (Nervous system disorders) | 2 (4)
Taste disturbance (dysgeusia) (Nervous system disorders) | 12 (25)
Urinary retention (Renal and urinary disorders) | 2 (2)
Urticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 2 (4)
Voice changes/stridor/larynx (e.g., hoarseness, loss of voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 7 (9)
Weight loss (Investigations) | 13 (17)
Wound-infectious (Infections and infestations) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes